CLINICAL TRIAL: NCT05847114
Title: Investigation of the Effects of Stress Ball Practice on Patients Anxiety, Pain and Vital Signs During Cataract Surgery
Brief Title: Evaluation of the Effectiveness of Stress Ball Practice During Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Seda Cansu Yenigun, Student, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EGE-PhD-9319000443
Record Dates: First submitted 2023-04-04; First posted 2023-05-06 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cataract; Anxiety; Pain
Keywords: cataract; stress ball; anxiety; pain; vital signs
MeSH Terms: conditions — Cataract; Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stress Ball Group (Experimental): VAS-A, VAS, Spielberg Trait Anxiety Inventory was applied. Vital signs were evaluated before, during and after surgery. Stress balls were given to the patients in addition to the standard care protocol. Stress balls were used for 15 minutes during the operation, by placing the patient in both hands, counting from one to five, and tightening and loosening twice.
  Interventions: Other: Stres ball
- Control Group (No Intervention): Patients in the control group will not undergo any intervention other than the standard care protocol.

INTERVENTIONS:
Other: Stres ball — Stress ball compression for 15 minutes during surgery
  Arms: Stress Ball Group

SUMMARY:
Cataract surgery is one of the most commonly performed and reliable surgeries among eye diseases. While cataract surgeries were performed under general or local anesthesia in previous years, they are now performed topically. Despite providing conscious sedation with agents such as benzodiazepines and opioids before and during surgery, patients experience pain, anxiety, and discomfort during the surgical procedure.

One of the non-pharmacological methods used to relieve acute pain during surgical intervention is stress ball. It is also used to reduce pain and anxiety and increase patient comfort. The stress ball suppresses most of the nerves and muscles directly connected to the brain around the wrist and hand, stimulating nerve and muscle activity. This mechanism reduces the release of stress hormones, regulates blood pressure by providing relaxation and relief, and helps reduce anxiety and acute stress.

When literature is examined, it is seen that stress ball application is effective on patients' pain, anxiety, and vital signs; however, no randomized controlled study has been found in which stress ball application was performed during cataract surgery. This study was planned to investigate the effect of stress ball application during cataract surgery on patients' anxiety, pain, and vital signs.

DETAILED DESCRIPTION:
After obtaining the permission of the ethics committee and institution of the study, the researcher will go to the clinic and introduce herself to the patient who is hospitalized for cataract surgery and explain the purpose of the research. Informed consent will be obtained from patients willing to participate in the study. The data on the socio-demographic characteristics of the patients in the patient introduction form will be interviewed face-to-face with the patient, and the data on the clinical features of the patients will be recorded from the patient file. Data will begin to be collected from the first patient who will go to surgery. Systolic-diastolic blood pressure, heart rate, respiration, O2 saturation will be measured and recorded 5-10 minutes before the surgery. Pain levels with VAS, anxiety levels with VAS-A and Spielberg Trait Anxiety Scale will be checked. According to the randomization, the patient in the stress ball group will first be given the stress balls in both palms by the researcher, and they will be asked to count from one to five and squeeze them twice. The patient will be shown to use stress balls for 15 minutes during the surgery and will be applied. The patient will be explained to use the stress balls for 15 minutes during the surgery. When the 15 minutes are up, the patient will be informed by the researcher and the patient will be able to let go of the stress balls. No intervention will be performed on the patient in the control group. The first patient will go to the operating room. After the patient goes to the operating table and the preparation for the surgery is completed, the patients in the stress ball group will practice the stress balls for 15 minutes. No intervention will be performed on the patient in the control group. At the 15th minute of the operation, a scale will be applied to all patient groups to determine the level of pain with VAS and anxiety level with VAS-A, and systolic-diastolic blood pressure, heart rate, and O2 saturation will be measured and recorded. At the end of the cataract surgery, the patient will be transferred to the service. The patient who is transferred to the service will be rested. The patient's systolic-diastolic blood pressure, heart rate, O2 saturation will be measured and recorded after 10 minutes. In addition, a scale will be applied to the patient to determine the pain level with VAS and the level of anxiety with VAS-A. No intervention will be made to the control group patients, and the routine care protocol of the clinic will be applied.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* Absence of hearing and perception problems,
* Having no physical problems to squeeze a stress ball,
* First time cataract surgery.

Exclusion Criteria:

* Using any analgesic or anxiolytic before surgery,
* Conversion of topical anesthesia to general anesthesia during surgery,
* Having a psychiatric disorder
* Uncontrolled hypertension in the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult, older adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Pain (Visual Analog Scale) | 15 minutes before surgery
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Pain (Visual Analog Scale) | During surgery
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Pain (Visual Analog Scale) | 10 minutes after surgery
  Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no pain and "10" means the most severe pain.
  The patient marks the intensity of pain he feels on the ruler. If the marked value is between 1-4, it indicates mild pain, between 5-6 indicates moderate pain, and between 7-10 indicates severe pain.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Anxiety (Visual Analog Scale-Anxiety) | 15 minutes before surgery, during surgery and 10 minutes after surgery
  Patients' anxiety will be evaluated (0-10 point). Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no anxiety and "10" means the most severe anxiety.
  In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
State-Trait Anxiety Inventory (STAI-II) | 15 minutes before surgery
  STAI-II is a well-researched clinical tool for evaluating the tendency towards anxiety. A cut-off point of 39-40 typically indicates clinically significant symptoms of a state of anxiety.
Vital signs | 15 minutes before surgery, during surgery and 10 minutes after surgery
  In the measurement of vital signs of individuals, devices that measure digital blood pressure and pulse, O2 saturation will be used by applying the necessary hygiene rules at patient transitions.The respiratory rate will also be checked.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Ege Üniversitesi Hemşirelik Fakültesi Bornova/İZMİR, Turkey (Türkiye)